CLINICAL TRIAL: NCT02902185
Title: Efficacy of the Histone Deacetylase Inhibitor Chidamide in Combination With Antiretroviral Therapy for Reactivation of the Latent HIV-1 Reservoir:a Randomized Controlled Clinical Trial
Brief Title: Chidamide in Combination With ART for Reactivation of the Latent HIV-1 Reservoir
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Chipscreen Biosciences, Ltd. (Industry); Zhejiang University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yongtao Sun, MD, PhD, Director of Department of Infectious Diseases, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016TD-Chidamide RCT
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Chronic HIV Infections
Keywords: Chidamide; Histone Deacetylase Inhibitor; HIV-1 Reservoir; Chronic HIV infections; HIV Eradication; Antiretroviral Therapy
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide (Experimental): Chidamide will be administrated 10mg each time, twice a week, interval not less than 3 days for 12 weeks.
  Interventions: Drug: ART plus Chidamide
- Placebo-controlled (Placebo Comparator): Placebo with the same taste and appearance like Chidamide will be administrated 10mg each time, twice a week, interval not less than 3 days for 12 weeks.
  Interventions: Drug: ART plus Placebo

INTERVENTIONS:
Drug: ART plus Chidamide — Chidamide will be administrated 10mg each time, twice a week, interval not less than 3 days for 12 weeks.Antiretroviral therapy will be kept during entire study.
  Arms: Chidamide
Drug: ART plus Placebo — Placebo will be administrated 10mg each time, twice a week, interval not less than 3 days for 12 weeks.Antiretroviral therapy will be kept during entire study.
  Arms: Placebo-controlled

SUMMARY:
HIV replication can be effectively suppressed and acquired immunodeficiency syndrome(AIDS) can be prevented with highly active antiretroviral therapy (HAART). However, HIV-infected people must remain on treatment continuously to avoid viral rebound and progression to AIDS. HIV persistence is thought to stem primarily from the presence of integrated copies of the proviral genome within long-lived cells. Because active viral gene expression causes cell death due to viral cytopathic effects and the immune response, long-lived cells likely harbor transcriptionally silent, latent provirus. HIV-1 persistence in long-lived cellular reservoirs remains a major barrier to a cure. HDACi have the potential to activate ("Kick") these latently infected cells. This will make the HIV infected cells visible to the immune system; the immune response and antiretrovirals(ARVs) will be able to attack and eliminate ("Kill") the infected cells. This study is subsequent to our NCT02513901. The purpose of this study is to verify the efficacy of multi-dose Chidamide in combination with antiretroviral therapy in HIV-infected adults with suppressed viral load in a randomized controlled clinical trial.

DETAILED DESCRIPTION:
Sixty participants will be recruited and stratified by their CD4 cell count(30 for <500 cells/μL and 30 for ≥500 cells/μL). Each layer was 1:1 randomly divided into Chidamide group or Placebo-controlled group.Chidamide and Placebo will be administrated 10mg each time, twice a week, interval not less than 3 days. Chidamide and Placebo intervention will last 12 consecutive weeks. All participants will keep their antiretroviral therapy during this study.

This study will last for 96 weeks, involving 16 study visits(Screening, Week 0, 2, 4, 8, 12, 14, 16, 20, 24, 36, 48, 60, 72, 84, 96) for every participant. At the screening visit, participants will give a medical history and will undergo a physical exam; blood samples will be collected. If participants agree, their blood samples may be stored for future research.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Currently receiving cART and having received cART for a minimum of 24 months, HIV-1 plasma RNA <20 copies/mL for at least 1.5 year (excluding viral load blips)
* CD4 T cell count >350 cells/mm3
* Able, willing to give written informed consent and to adhere to therapy and to comply with time requirements for study visits and evaluations
* Adequate vascular access for leukapheresis

Exclusion Criteria:

* Acute HIV-1 infection
* Received blood transfusions or hematopoetic growth factors within 3 months receipt of compounds with HDAC inhibitor-like activity, such as valproic acid within the last 1 month. Potential participants may enroll after a 30-day washout period.
* Any significant acute medical illness in the past 8 weeks
* Any evidence of an active AIDS-defining opportunistic infection
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood
* Patient has the following laboratory values within 3 weeks before starting the investigational drug

  1. Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  2. Serum total bilirubin ≥1.5 ULN
  3. Serum creatinine levels ≥1.5 x ULN, or calculated creatinine clearance ≤60 ml/min
  4. Platelet count ≤100 x109/L
  5. Absolute neutrophil count ≤1.5x109/L
  6. Serum potassium, magnesium, phosphorus outside normal limits
  7. Total calcium (corrected for serum albumin) or ionized calcium ≤lower normal limits
* A personal history of clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for Torsades de pointes (e.g. heart failure)
* History of malignancy or transplantation, including skin cancers or Kaposi sarcoma
* History of diabetes mellitus
* Known hypersensitivity to the components of chidamide or its analogues
* Pregnancy or breast feeding, or expecting to father children within the projected duration of the study
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in HIV transcription measured as cell associated HIV-1 RNA (copies per 10E6 PBMCs) | Measured on week 0, 2, 4, 8, 12, 14, 16, 24
Change in HIV production measured as plasma HIV RNA (by Roche COMBAS TaqMan HIV-1 Test version 2.0) | Measured on week 0, 2, 4, 8, 12, 14, 16, 24, 36, 48, 60, 72, 84, 96
Change in HIV-1 reservoir size measured in PBMCs by Total HIV-1 DNA(copies per 10E6 PBMCs) | Measured on week 0, 2, 4, 8, 12, 14, 16, 24, 36, 48, 60, 72, 84, 96

SECONDARY OUTCOMES:
Safety and tolerability evaluation as measured by adverse events (AE), adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR), serious unexpected adverse reactions (SUSAR) | Measured through 96 weeks
Cell surface markers of immune activation and immune checkpoints and so on | Measured on week 0, 2, 4, 8, 12, 14, 16, 24, 36, 48, 60, 72, 84, 96
Plasma inflammatory biomarkers | Measured on week 0, 4, 8, 12, 16, 24, 48, 72, 96

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Department of Infectious Diseases, Tangdu Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
We do not have data share plan because of participants' privacy.